CLINICAL TRIAL: NCT01116882
Title: A Randomized Trial to Compare Percutaneous Coronary Intervention Between Massachusetts Hospitals With Cardiac Surgery-On-Site and Community Hospitals Without Cardiac Surgery-On-Site
Brief Title: Percutaneous Coronary Intervention (PCI) Outcomes in Community Versus Tertiary Settings
Acronym: MASS COMM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Baim Institute for Clinical Research (Other)
Collaborators: Brockton Hospital (Other); Good Samaritan Hospital Medical Center, New York (Other); Norwood Hospital (Other); Holy Family Hospital, Methuen, MA (Other); Lawrence General Hospital (Unknown); Lowell General Hospital (Other); Melrose Wakefield Hospital (Unknown); Metro West Medical Center (Other); Saints Memorial Medical Center (Unknown); South Shore Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: DPH00
Record Dates: First submitted 2010-04-29; First posted 2010-05-05 (Estimated); Results first posted 2014-07-08 (Estimated); Last update posted 2015-04-07 (Estimated); Status verified 2015-03

CONDITIONS: Coronary Artery Diseases
Keywords: PCI; heart disease; ischemic heart disease
MeSH Terms: conditions — Coronary Artery Disease; Heart Diseases; Myocardial Ischemia

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- SOS (Active Comparator): Patients randomized to the SOS arm are transferred to tertiary hospitals for their PCI procedure.
  Interventions: Procedure: PCI
- Non-SOS (Experimental): Patients in the non-SOS arm are randomized to stay at the community hospitals for their PCI procedure.
  Interventions: Procedure: PCI

INTERVENTIONS:
Procedure: PCI

SUMMARY:
The primary objective of the trial is to compare the acute safety and long term outcomes between hospitals with cardiac surgery on-site (SOS hospitals) and hospitals without cardiac surgery on-site (non-SOS hospitals) for patients with ischemic heart disease treated with elective percutaneous coronary intervention (PCI) (stable angina, acute coronary syndrome, or non-Q wave MI) presenting to non-SOS hospitals.

DETAILED DESCRIPTION:
The MASS COMM trial is a prospective, multi-center, randomized, controlled two-arm trial of PCI performed at non-SOS hospitals (non-SOS-PCI arm) versus PCI performed at SOS hospitals (SOS-PCI arm). The trial is designed to reject the null-hypothesis of inferiority, and thereby show the non-inferiority of the non-SOS-PCI arm to the SOS-PCI arm.

Specifically, 3690 subjects will be enrolled in a multi-center, randomized, controlled trial (RCT), in which eligible subjects will be consented and randomized in a 3:1 ratio at the non-SOS hospitals for PCI to be performed at either the enrolling non-SOS hospital (3 chances out of 4) or a corresponding SOS hospital (1 chance out of 4).

ELIGIBILITY:
Inclusion Criteria:

1. Subject is at least 18 years old.
2. Subject requires single- or multi-vessel percutaneous coronary intervention (PCI) of de novo or restenotic target lesion (including in-stent restenotic lesions).
3. Subject's lesion(s) is (are) amenable to stent treatment with currently available FDA-approved bare metal or drug eluting stents.
4. Subject is an acceptable candidate for elective, urgent or emergency coronary artery bypass graft (CABG).
5. Subject has clinical evidence of ischemic heart disease in terms of a positive functional study, or documented symptoms.
6. Documented stable angina pectoris [Canadian Cardiovascular Society Classification (CCS) 1, 2, 3, or 4], unstable angina pectoris with documented ischemia (Braunwald Class IB-C, IIB-C, or IIIB-C), non-ST segment elevation myocardial infarction, or documented silent ischemia.
7. Subject is willing and able to undergo percutaneous intervention at SOS hospital, if randomized to SOS study arm.
8. Subject and the treating physician agree that the subject will comply with all follow-up evaluations.
9. Subject has been informed of the nature of the study and agrees to its provisions and has provided written informed consent as approved by the Institutional Review Board/Ethics Committee of the respective clinical site.
10. The target lesion(s) is (are) de novo or restenotic (including in-stent restenotic) native coronary artery lesion(s) with greater than 50 and less than 100% stenosis (visual estimate), or the target lesion is an acute (less than 1 month) total occlusion as evidenced by clinical symptoms.
11. Target lesions(s) is (are) located in an infarct (if not treated with primary PCI) or non-infarct-related artery with a 70% or greater stenosis (by visual estimate) more than 72 hours following the ST segment elevation myocardial infarction (STEMI).

Lesions treated with PCI more than 72 hours following STEMI would be subject to the same protocol inclusion/exclusion criteria listed above and below with the exception that a target lesion of 70% or greater stenosis may be treated with or without symptoms or abnormal stress test).

Exclusion Criteria:

1. The patient is pregnant or breastfeeding.
2. Evidence of STEMI within 72 hours of the intended treatment on infarct related or non-infarct related artery.
3. Cardiogenic shock on presentation or during current hospitalization.
4. Left ventricular ejection fraction less than 20%.
5. Known allergies to: aspirin, clopidogrel (Plavix) and ticlopidine (Ticlid), heparin, bivalirudin, stainless steel, or contrast agent (which cannot be adequately premedicated).
6. A platelet count less than 75,000 cells/mm3 or greater than 700,000 cells/mm3 or a WBC less than 3,000 cells/mm3.
7. Acute or chronic renal dysfunction (creatinine greater than 2.5 mg/dl or less than 150µmol/L).
8. Subject is currently participating in an investigational drug or device study that has not completed the primary endpoint or that clinically interferes with the current study endpoints. (Note: Trials requiring extended follow-up for products that were investigational, but have since become commercially available, are not considered investigational trials).
9. Prior participation in this study.
10. Within 30 days prior to the index study procedure, the subject has undergone a previous coronary interventional procedure of any kind. Note: This exclusion criterion does not apply to post-STEMI patients.
11. Stroke or transient ischemic attack within the prior 3 months.
12. Active peptic ulcer or upper gastrointestinal bleeding within the prior 3 months.
13. Subject has active sepsis.
14. Unprotected left main coronary artery disease (stenosis greater than 50%).
15. In the investigator's opinion, subject has a co-morbid condition(s) that could limit the life expectancy to less than one year, or limit the subject's ability to participate in the study or comply with follow-up requirements or impact the scientific integrity of the study.
16. Subject has normal or insignificant coronaries (i.e. coronary lesion(s) less than 50% stenosis).
17. Any target vessel has evidence of:

    * excessive thrombus (e.g. requires target vessel thrombectomy)
    * tortuousity (greater than 60 degree angle) that makes it unsuitable for proper stent delivery and deployment,
    * heavy calcification.
18. Any target lesion requires treatment with a device other than percutaneous transluminal coronary angioplasty (PTCA) prior to stent placement (e.g. but not limited to, directional coronary atherectomy, excimer laser, rotational atherectomy, etc.).
19. Any lesion that is located in a saphenous vein graft, however, lesions located within the native vessel but accessed through the graft are eligible.
20. The target vessel is in a "last remaining" epicardial vessel (e.g. greater than 2 non-target epicardial vessels and the bypass grafts to these territories [if present] are totally occluded).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3691 (Actual)
Dates: Start 2006-06; Primary Completion 2012-06 (Actual); Study Completion 2012-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Alice K Jacobs, MD, Principal Investigator — Boston University School of Medicine , Boston Medical Center; Sharon-Lise Normand, Ph.D., Principal Investigator — Harvard Medical School (HMS and HSDM); Laura Mauri, M.D., Principal Investigator — Brigham and Women's Hospital
Locations (17):
- United States (17):
  - Tufts New England Medical Center, Boston, Massachusetts
  - Massachusetts General Hospital, Boston, Massachusetts
  - Boston University Medical Center, Boston, Massachusetts
  - Brigham and Women's Hospital, Boston, Massachusetts
  - Beth Israel Deaconnes Medical Center, Boston, Massachusetts
  - Caritas St. Elizabeth's Hospital, Brighton, Massachusetts
  - Brockton Hospital, Brockton, Massachusetts
  - Caritas Good Samaritan Medical Center, Brockton, Massachusetts
  - Lahey Clinic, Burlington, Massachusetts
  - Metrowest Medical Center, Framingham, Massachusetts
  - Lawrence General Hospital, Haverhill, Massachusetts
  - Saints Memorial Medical Center, Lowell, Massachusetts
  - Lowell General Hospital, Lowell, Massachusetts
  - Melrose Wakefield Hospital, Melrose, Massachusetts
  - Caritas Holy Family Hospital, Methuen, Massachusetts
  - Caritas Norwood Hospital, Norwood, Massachusetts
  - South Shore Hospital, Weymouth, Massachusetts

REFERENCES:
- [Derived] Jacobs AK, Normand SL, Massaro JM, Cutlip DE, Carrozza JP Jr, Marks AD, Murphy N, Romm IK, Biondolillo M, Mauri L; MASS COMM Investigators. Nonemergency PCI at hospitals with or without on-site cardiac surgery. N Engl J Med. 2013 Apr 18;368(16):1498-508. doi: 10.1056/NEJMoa1300610. Epub 2013 Mar 11. PMID 23477625
- [Derived] Mauri L, Normand SL, Pencina M, Cutlip DE, Jeon C, Dreyer P, Kuntz RE, Baim DS, Jacobs AK. Rationale and design of the MASS COMM trial: A randomized trial to compare percutaneous coronary intervention between MASSachusetts hospitals with cardiac surgery on-site and COMMunity hospitals without cardiac surgery on-site. Am Heart J. 2011 Nov;162(5):826-31. doi: 10.1016/j.ahj.2011.08.018. PMID 22093197

RESULTS

PARTICIPANT FLOW:
Groups:
- PCI at a Hospital Without On-site Cardiac Surgery: Assigned to PCI at a hospital without on-site cardiac surgery
- PCI at Hospital With On-Site Cardiac Surgery: Assigned to PCI at a hospital with on-site cardiac surgery
Period: 30-day
Arm/Group | PCI at a Hospital Without On-site Cardiac Surgery | PCI at Hospital With On-Site Cardiac Surgery
Started | 2774 | 917
Completed | 2706 | 886
Not Completed | 68 | 31
Not completed — Lost to Follow-up | 50 | 21
Not completed — Withdrawal by Subject | 2 | 4
Not completed — Other Reasons | 16 | 6
Period: 12-month
Arm/Group | PCI at a Hospital Without On-site Cardiac Surgery | PCI at Hospital With On-Site Cardiac Surgery
Started | 2706 | 886
Completed | 2439 | 787
Not Completed | 267 | 99
Not completed — Lost to Follow-up | 111 | 42
Not completed — Other Reasons | 151 | 49
Not completed — Withdrawal by Subject | 5 | 8

BASELINE CHARACTERISTICS:
Groups:
- PCI at Hospitals Without On-Site Cardiac Surgery: Assigned to PCI at a hospital without on-site cardiac surgery
- Total: Total of all reporting groups
Arm/Group | PCI at Hospitals Without On-Site Cardiac Surgery | PCI at Hospital With On-Site Cardiac Surgery | Total
Number analyzed (Participants) | 2774 | 917 | 3691
Age, Continuous [Mean (Standard Deviation); unit: years] | 64.71 (11.84) | 64.16 (11.81) | 64.57 (11.83)
Sex/Gender, Customized [Number; unit: participants]
  Female | 883 | 308 | 1191
  Male | 1891 | 609 | 2500
Race/Ethnicity, Customized [Number; unit: participants]
  White | 2526 | 852 | 3378
  Black | 51 | 9 | 60
  Hispanic | 117 | 35 | 152
  Other | 80 | 21 | 101

OUTCOME MEASURES:

1. Primary Outcome: 30-day Composite Major Adverse Cardiac Event (MACE)
Time Frame: 30 days
Population: The denominator for MACE at 30 days is defined as patients who either had MACE to 30d or had follow up of at least 23 days.
Measure: Number; unit: participants
Arm/Group | PCI at Hospitals Without On-Site Cardiac Surgery | PCI at Hospital With On-Site Cardiac Surgery
Number analyzed (Participants) | 2706 | 886
participants | 256 | 83

2. Primary Outcome: 12-month Composite Major Adverse Cardiac Event (MACE)
Time Frame: 12 month
Measure: Number; unit: participants
Arm/Group | PCI at Hospitals Without On-Site Cardiac Surgery | PCI at Hospital With On-Site Cardiac Surgery
Number analyzed (Participants) | 2439 | 787
participants | 421 | 140

3. Secondary Outcome: All Cause Mortality at 30 Days
Time Frame: 30 days
Population: The denominator for MACE at 30 days is defined as patients who either died to 30d or had follow up of at least 23 days.
Measure: Number; unit: participants
Arm/Group | PCI at Hospitals Without On-Site Cardiac Surgery | PCI at Hospital With On-Site Cardiac Surgery
Number analyzed (Participants) | 2708 | 885
participants | 18 | 3

4. Secondary Outcome: Ischemia-driven Target Lesion Revascularization
Time Frame: 30 days
Measure: Number; unit: participants
Arm/Group | PCI at Hospitals Without On-Site Cardiac Surgery | PCI at Hospital With On-Site Cardiac Surgery
Number analyzed (Participants) | 2689 | 882
participants | 36 | 12

5. Secondary Outcome: Ischemia-driven Target Lesion Revascularization
Time Frame: 12 months
Measure: Number; unit: participants
Arm/Group | PCI at Hospitals Without On-Site Cardiac Surgery | PCI at Hospital With On-Site Cardiac Surgery
Number analyzed (Participants) | 2364 | 766
participants | 117 | 38

6. Secondary Outcome: Rate of Stent Thrombosis
Time Frame: 12 months
Measure: Number; unit: participants
Arm/Group | PCI at Hospitals Without On-Site Cardiac Surgery | PCI at Hospital With On-Site Cardiac Surgery
Number analyzed (Participants) | 2364 | 771
participants | 27 | 16

7. Secondary Outcome: Any Repeat Revascularization
Time Frame: 12 months
Measure: Number; unit: participants
Arm/Group | PCI at Hospitals Without On-Site Cardiac Surgery | PCI at Hospital With On-Site Cardiac Surgery
Number analyzed (Participants) | 2372 | 769
participants | 202 | 76

8. Secondary Outcome: Emergency or Urgent Revascularization
Time Frame: 30 days
Population: The denominator for emergency or urgent revascularization at 30 days is defined as patients who either had the event to 30d or had follow up of at least 23 days.
Measure: Number; unit: participants
Arm/Group | PCI at Hospitals Without On-Site Cardiac Surgery | PCI at Hospital With On-Site Cardiac Surgery
Number analyzed (Participants) | 2774 | 917
participants | 7 | 2

9. Secondary Outcome: Procedural Success
Description: Procedural success is defined as residual stenosis of the target lesion of less than 20%
Time Frame: Post-Procedure
Measure: Number; unit: participants
Groups:
- PCI at Hospitals Without On-Site Cardiac Surgery: Assigned to PCI at a hospital without on-site cardiac surgery in the angiographic cohort
- PCI at Hospital With On-Site Cardiac Surgery: Assigned to PCI at a hospital with on-site cardiac surgery in the angiographic cohort
Arm/Group | PCI at Hospitals Without On-Site Cardiac Surgery | PCI at Hospital With On-Site Cardiac Surgery
Number analyzed (Participants) | 289 | 87
participants | 235 | 65

10. Secondary Outcome: Major Vascular Complications
Time Frame: 30 days
Measure: Number; unit: participants
Arm/Group | PCI at Hospitals Without On-Site Cardiac Surgery | PCI at Hospital With On-Site Cardiac Surgery
Number analyzed (Participants) | 2687 | 882
participants | 41 | 13

11. Secondary Outcome: Complete Revascularization
Description: Complete revascularization was defined as the successful treatment, according to the criteria of procedural success, of all epicardial vessels with more than 70% and less than 100% stenosis.
Time Frame: Post-Procedure
Measure: Number; unit: participants
Arm/Group | PCI at Hospitals Without On-Site Cardiac Surgery | PCI at Hospital With On-Site Cardiac Surgery
Number analyzed (Participants) | 289 | 87
participants | 174 | 52

12. Secondary Outcome: Met Indication Criteria for PCI
Description: Included here are the number of treated lesions that met the class I or II recommendations for anatomical indications for PCI, according to the PCI guidelines fo the American College of Cardiology Foundation-American Heart Association-Society for Cardiovascular Angiography and Interventions.
Time Frame: Post-Procedure
Measure: Number; unit: lesions
Units Other Than Participants: Lesions
Arm/Group | PCI at Hospitals Without On-Site Cardiac Surgery | PCI at Hospital With On-Site Cardiac Surgery
Number analyzed (Participants) | 289 | 87
Number analyzed (Lesions) | 392 | 106
lesions | 369 | 97

13. Secondary Outcome: All Cause Mortality at 12 Months
Time Frame: 12 months
Measure: Number; unit: participants
Arm/Group | PCI at Hospitals Without On-Site Cardiac Surgery | PCI at Hospital With On-Site Cardiac Surgery
Number analyzed (Participants) | 2424 | 785
participants | 56 | 19

14. Secondary Outcome: Ischemia-driven Target Vessel Revascularization
Time Frame: 30 days
Measure: Number; unit: participants
Arm/Group | PCI at Hospitals Without On-Site Cardiac Surgery | PCI at Hospital With On-Site Cardiac Surgery
Number analyzed (Participants) | 2689 | 882
participants | 41 | 13

15. Secondary Outcome: Ischemia-driven Target Vessel Revascularization
Time Frame: 12 months
Measure: Number; unit: participants
Arm/Group | PCI at Hospitals Without On-Site Cardiac Surgery | PCI at Hospital With On-Site Cardiac Surgery
Number analyzed (Participants) | 2366 | 766
participants | 133 | 41

16. Secondary Outcome: Rate of Stent Thrombosis
Time Frame: 30 days
Measure: Number; unit: participants
Arm/Group | PCI at Hospitals Without On-Site Cardiac Surgery | PCI at Hospital With On-Site Cardiac Surgery
Number analyzed (Participants) | 2695 | 883
participants | 16 | 7

17. Secondary Outcome: Any Repeat Revascularization
Time Frame: 30 days
Population: The denominator for any repeat revascularization at 30 days is defined as patients who either had the event to 30d or had follow up of at least 23 days.
Measure: Number; unit: participants
Arm/Group | PCI at Hospitals Without On-Site Cardiac Surgery | PCI at Hospital With On-Site Cardiac Surgery
Number analyzed (Participants) | 2689 | 883
participants | 73 | 31

ADVERSE EVENTS:
Description: Serious and other adverse events were not collected in this study.
Groups:
- Non-Surgery-On-Site (Non-SOS): Patients in the non-SOS arm are randomized to stay at the community hospitals for their PCI procedure.
- Surgery-On-Site (SOS): Patients randomized to the SOS arm are transferred to tertiary hospitals for their PCI procedure.
Arm/Group | Non-Surgery-On-Site (Non-SOS) | Surgery-On-Site (SOS)
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No